CLINICAL TRIAL: NCT04227873
Title: Sleep and Cognition After Ambulatory Hip and Knee Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Kehlet, Henrik, M.D., Ph.D. (Individual); Nicolai Bang Foss (Unknown); Poul Jenum (Unknown); Anders Troelsen (Unknown); Kirill Gromov (Unknown); Mette Grentoft (Unknown); Henning Piilgaard Hansen (Unknown)
Responsible Party: Principal Investigator, Alexandre Garioud, Principal investigator, Hvidovre University Hospital
Other Study IDs: HVH01
Record Dates: First submitted 2019-12-12; First posted 2020-01-14 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Sleep Disturbance; Delirium; Arthroplasty Complications
MeSH Terms: conditions — Parasomnias; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sleep and rest are key elements in postoperative rehabilitation and recovery. There are complex relations between major surgery, sleep disturbance and complications. Major surgery leeds to severe postoperative sleep disturbances, initially reducing REM sleep time and disturbing the remaining sleep stages. Major surgery is again a risk factor for postoperative delirium and other cognitive impairment. The underlying mechanisms includes pain, opioid medication, sleep disturbances and neuroinflammation, along with external factors as noise during hospitalisation. The physiologic stress from sleep disturbances and sleep deprivation is associated with blood-brain barrier impairment, inflammation, decreased restitution, altered nociceptive function. Likewise, undiagnosed and untreated sleep apnea is a risk for postoperative complications and is itself affected by anesthesia and some analgesics (i.a. opioids).

Fast-track surgery development has led to restitution period shortening, optimized pain management reducing opioid use, postoperative inflammatory stress response reduction and less delirium. Evolution of hip and knee arthroplasty(THA/TKA), organisation, optimized pain management and pharmacologic modification of inflammatory response by high dose steroid has permitted to perform these surgeries in an outpatient setting.

Previous studies of fast-track THA/TKA using multimodal opioid-sparring analgesia, however neither using high dose steroids nor in an out patient setting, have demonstrated REM sleep period reduction from a normal range of 18% preoperatively to 1% postoperatively. However, changes in sleep architecture after THA/TKA in at setting attempting to minimise abnormal sleep by means of ambulatory surgery added to perioperative reduction of inflammatory response to surgery, pain and opioid use by high dose steroid, haven't been studied.

The purpose of this study is to investigate how much an optimized ambulatory THA/TKA , reducing pain and inflammatory response to surgery and opioid use by high doses steroid can conserve the preoperative sleep architecture.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification I or II
* Scheduled hospital discharge same day after surgery
* Adult person following the patient 24 hours at the patients habitation
* Informed consent and signature.
* Patient speaks and understands Danish

Exclusion Criteria:

* Hospital discharge later than same day after surgery
* No consent form patient
* Alcohol or drug abuse
* Anxiolytic og antipsychotic treatment
* Preoperative opioid treatment
* Soporific treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 16 adult attending scheduled hip or knee arthroplasty in an ambulatory fast-track setting with spinal anesthesia corresponding to the above mentioned inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Changes in postoperative REM sleep time compared to preoperative | One night 2 to 4 night preoperatively, and the first and second postoperative night.
  Polysomnography

SECONDARY OUTCOMES:
Changes Remaining sleep stages and sleep variables (i.a. apnea) | One night 2 to 4 night preoperatively, and the first and second postoperative night.
  Polysomnography
Presence and severity of postoperative delirium compared to preoperative | One night 2 to 4 night preoperatively, and after the second postoperative night.
  Confusion Assessement Method-Severity (CAM-S). High scores, better outcome.
Presence and severity of postoperative cognitive impairment compared to preoperative | One night 2 to 4 night preoperatively, and after the second postoperative night.
  Mini Mental State Examination (MMSE), High scores, better outcome.

OTHER OUTCOMES:
Subjective measurement of tiredness | One night 2 to 4 night preoperatively, and after the second postoperative night.
  questionnaire. Better sleep, better outcome.
Subjective measurement of sleep quality | One night 2 to 4 night preoperatively, and after the second postoperative night.
  Pittsburgh Sleep Quality Index. Lower score, better outcome.
Changes in preoperative inflammatory marker level (CRP) compared to postoperative. | One night 2 to 4 night preoperatively, and after the second postoperative night.
  Blod samples
Subjective measurements of pain at rest and after mobilisation. | Immediately after surgery, and after the first and second postoperative night.
  questionnaire. Visual Analogue Scale(VAS). Lower score, better outcome.
Registration of opioid use. | Immediately after surgery, and after the first and second postoperative night.
  questionnaire. Less opioid use, better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Kehlet, Dr.med,Phd, Study Director — Rigshospitalet, Denmark
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aldecoa C, Bettelli G, Bilotta F, Sanders RD, Audisio R, Borozdina A, Cherubini A, Jones C, Kehlet H, MacLullich A, Radtke F, Riese F, Slooter AJ, Veyckemans F, Kramer S, Neuner B, Weiss B, Spies CD. European Society of Anaesthesiology evidence-based and consensus-based guideline on postoperative delirium. Eur J Anaesthesiol. 2017 Apr;34(4):192-214. doi: 10.1097/EJA.0000000000000594. PMID 28187050
- [Background] Inouye SK, Kosar CM, Tommet D, Schmitt EM, Puelle MR, Saczynski JS, Marcantonio ER, Jones RN. The CAM-S: development and validation of a new scoring system for delirium severity in 2 cohorts. Ann Intern Med. 2014 Apr 15;160(8):526-533. doi: 10.7326/M13-1927. PMID 24733193
- [Background] Keats AS. The ASA classification of physical status--a recapitulation. Anesthesiology. 1978 Oct;49(4):233-6. doi: 10.1097/00000542-197810000-00001. No abstract available. PMID 697075
- [Result] Krenk L, Rasmussen LS, Kehlet H. New insights into the pathophysiology of postoperative cognitive dysfunction. Acta Anaesthesiol Scand. 2010 Sep;54(8):951-6. doi: 10.1111/j.1399-6576.2010.02268.x. Epub 2010 Jul 12. PMID 20626359
- [Result] Krenk L, Jennum P, Kehlet H. Postoperative sleep disturbances after zolpidem treatment in fast-track hip and knee replacement. J Clin Sleep Med. 2014 Mar 15;10(3):321-6. doi: 10.5664/jcsm.3540. PMID 24634631
- [Result] Krenk L, Jennum P, Kehlet H. Sleep disturbances after fast-track hip and knee arthroplasty. Br J Anaesth. 2012 Nov;109(5):769-75. doi: 10.1093/bja/aes252. Epub 2012 Jul 24. PMID 22831887
- [Result] Riedel B, Browne K, Silbert B. Cerebral protection: inflammation, endothelial dysfunction, and postoperative cognitive dysfunction. Curr Opin Anaesthesiol. 2014 Feb;27(1):89-97. doi: 10.1097/ACO.0000000000000032. PMID 24300462
- [Result] Ni P, Dong H, Zhou Q, Wang Y, Sun M, Qian Y, Sun J. Preoperative Sleep Disturbance Exaggerates Surgery-Induced Neuroinflammation and Neuronal Damage in Aged Mice. Mediators Inflamm. 2019 Mar 18;2019:8301725. doi: 10.1155/2019/8301725. eCollection 2019. PMID 31011286
- [Result] He J, Hsuchou H, He Y, Kastin AJ, Wang Y, Pan W. Sleep restriction impairs blood-brain barrier function. J Neurosci. 2014 Oct 29;34(44):14697-706. doi: 10.1523/JNEUROSCI.2111-14.2014. PMID 25355222
- [Result] McMahon WR, Ftouni S, Drummond SPA, Maruff P, Lockley SW, Rajaratnam SMW, Anderson C. The wake maintenance zone shows task dependent changes in cognitive function following one night without sleep. Sleep. 2018 Oct 1;41(10). doi: 10.1093/sleep/zsy148. PMID 30169703
- [Result] de Raaff CAL, Gorter-Stam MAW, de Vries N, Sinha AC, Jaap Bonjer H, Chung F, Coblijn UK, Dahan A, van den Helder RS, Hilgevoord AAJ, Hillman DR, Margarson MP, Mattar SG, Mulier JP, Ravesloot MJL, Reiber BMM, van Rijswijk AS, Singh PM, Steenhuis R, Tenhagen M, Vanderveken OM, Verbraecken J, White DP, van der Wielen N, van Wagensveld BA. Perioperative management of obstructive sleep apnea in bariatric surgery: a consensus guideline. Surg Obes Relat Dis. 2017 Jul;13(7):1095-1109. doi: 10.1016/j.soard.2017.03.022. Epub 2017 Mar 30. PMID 28666588
- [Result] Kehlet H. Fast-track hip and knee arthroplasty. Lancet. 2013 May 11;381(9878):1600-2. doi: 10.1016/S0140-6736(13)61003-X. No abstract available. PMID 23663938
- [Result] Kehlet H, Lindberg-Larsen V. High-dose glucocorticoid before hip and knee arthroplasty: To use or not to use-that's the question. Acta Orthop. 2018 Oct;89(5):477-479. doi: 10.1080/17453674.2018.1475177. Epub 2018 May 21. No abstract available. PMID 29781366
- [Result] Krenk L, Rasmussen LS, Hansen TB, Bogo S, Soballe K, Kehlet H. Delirium after fast-track hip and knee arthroplasty. Br J Anaesth. 2012 Apr;108(4):607-11. doi: 10.1093/bja/aer493. Epub 2012 Jan 24. PMID 22277666
- [Result] Gromov K, Kjaersgaard-Andersen P, Revald P, Kehlet H, Husted H. Feasibility of outpatient total hip and knee arthroplasty in unselected patients. Acta Orthop. 2017 Oct;88(5):516-521. doi: 10.1080/17453674.2017.1314158. Epub 2017 Apr 20. PMID 28426262
- [Result] Stephansen JB, Olesen AN, Olsen M, Ambati A, Leary EB, Moore HE, Carrillo O, Lin L, Han F, Yan H, Sun YL, Dauvilliers Y, Scholz S, Barateau L, Hogl B, Stefani A, Hong SC, Kim TW, Pizza F, Plazzi G, Vandi S, Antelmi E, Perrin D, Kuna ST, Schweitzer PK, Kushida C, Peppard PE, Sorensen HBD, Jennum P, Mignot E. Neural network analysis of sleep stages enables efficient diagnosis of narcolepsy. Nat Commun. 2018 Dec 6;9(1):5229. doi: 10.1038/s41467-018-07229-3. PMID 30523329